CLINICAL TRIAL: NCT02380131
Title: Phase IV Multi-Institutional Randomized Trial of Capecitabine Plus Oxaliplatin With Herceptin in Patients With Potentially Resectable HER-2 Positive Gastric Cancer With Liver Metastasis
Brief Title: Perioperative Chemotherapy With Herceptin For Potentially Resectable HER-2 Positive Gastric Cancer With Liver Metastasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alien-Craft 0002
Record Dates: First submitted 2013-10-08; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: HER-2 Positive Gastric Cancer; Liver Metastasis
Keywords: XELOX; Herceptin; Potentially Resectable Gastric Cancer
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Herceptin (Experimental): drug: Oxaliplatin;Capecitabine;Herceptin A cycle:Capecitabine 2000mg/m2 D1-D14 q3wk、Oxaliplatin 130 mg/m2 D1 q3wk add and subtract. Herceptin 8mg/kg D1 q3wk for the first time,after Herceptin 6mg/kg D1 q3wk.Evaluation for every two cycles.Each of preoperative and postoperative chemotherapy was 3 cycles.
  To explore the effect of herceptin with chemotherapy for potentially resectable HER-2 positive gastric cancer with liver metastasis
  Interventions: Drug: Oxaliplatin plus Capecitabine; Drug: Herceptin

INTERVENTIONS:
Drug: Oxaliplatin plus Capecitabine — A cycle: Oxaliplatin 130 mg/m2 D1 q3wk.E Capecitabine 2000mg/m2 D1-D14 q3wk、valuation for every two cycles.
  Other Names: Oxaliplatin plus capecitabine other names:XELOX.
Drug: Herceptin — Herceptin 8mg/kg D1 q3wk for the first time,after Herceptin 6mg/kg D1 q3wk.Evaluation for every two cycles.Each of preoperative and postoperative chemotherapy was 3 cycles.
  Other Names: Trastuzumab

SUMMARY:
Stage I：preoperative therapy

* Capecitabine plus oxaliplatin with herceptin is superior to surgery alone for patients with potentially resectable HER-2 positive gastric cancer with liver metastasis; Stage II: Perioperative therapy
* Perioperative Capecitabine plus oxaliplatin with herceptin is superior to adjuvant Capecitabine plus oxaliplatin alone for patients with potentially resectable HER-2 positive gastric cancer with liver metastasis;

DETAILED DESCRIPTION:
The investigators assessed whether the addition of a perioperative regimen of XELOX regimen with herceptin to improves R0 resection rate and survival among patients with potentially resectable HER-2 positive gastric cancer with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathological tissue were gastric cancer by gastric and liver biopsy.

  2.Immunohistochemistry confirmed HER-2 (+)or FISH(+).

  3.gastric cancer with liver metastasis were not able to resectable lesions.

  4.Patients•had not received radiotherapy past and not other organ metastasis and peritoneal metastasis.

  5.ECOG performance status 0-1.

  6.Inadequate hematopoietic function： Hemoglobin≥90g/L; ANC≥1,500/mm3;Platelet≥100,000/mm3 7.Inadequate organ function which is defined as below: Total bilirubin≤1.5 pper limit of normal range (ULN); ALT / AST≤2.5 upper limit of normal range (ULN) (≤5.0 x ULN if hepatic metastasis); serum creatinine≤1.5 pper limit of normal range (ULN), Serum albumin≥30g/L.

  8.expectancy must be more than 3 months. 9.the random blood or urine pregnancy test in fertile woman must be the negative results in pregnancy test in 7 days.

  10.Patients for male and female used reliable contraception contraceptive method until the end of study 30 days later.

  11.The operation can complete the D2 operation(LNM≥15).

  12.LVEF≥50%

Exclusion Criteria:

* 1. Patients with other extrahepatic metastasis Include peritoneal metastasis.

  3. Patients with other malignancy in 5 years.

  4. Patients with peripheral nerve disease,two hydrogen pyrimidine dehydrogenase( DPD )deficiency,upper digestive tract obstruction or from malabsorption syndrome.

  5.Patients with hypertension failed to control, active bleeding, 3~4 proteinuria, heal the wound, romboembolism, heart failure, clinical symptoms of heart disease.

  6.Patients have obvious peripheral nervous system disorders,mental disorders and disorders of the central nervous system history.

  7.Patients have history of organ transplantation.

  8.Patients with any medical or psychiatric condition or disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study.

  9.Patients combined antitumor drug outside the research program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | within 3 weeks after surgery

OTHER OUTCOMES:
R0-resection rate | within 3 weeks after surgery
Overall survival (OS) | 2 years
The number of Participants with adverse events | 2 years
  Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Doctor, Principal Investigator — Hebei Medical University
Locations (1):
- Department of Internal Medicine-Oncology, Shijiazhuang, Hebei, China